CLINICAL TRIAL: NCT00535509
Title: Phase II Trial of Neoadjuvant[FEC100]/Cisplatin-Docetaxel ± Trastuzumab in Women With Over Expressed or Amplified Her2/Neu With Locally Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Dr. Naeem A. Chaudhri, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC #2061-048
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Cisplatin-Docetaxel ± Trastuzumab — Chemo & RT
Other: Cisplatin-Docetaxel ± Trastuzumab — Chemo & RT
Drug: Cisplatin-Docetaxel ± Trastuzumab — Chemo & RT

SUMMARY:
Phase II trial of Neoadjuvant [FEC100]/Cisplatin-Docetaxel ± Trastuzumab in women with over expressed or amplified Her2/Neu with Locally advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced breast cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | overall

CONTACTS AND LOCATIONS:
Overall Officials: Taher Twegieri, MD, Principal Investigator — KFSH&RC; Dahish Ajarim, MD, Study Director — KFSH&RC